CLINICAL TRIAL: NCT04271566
Title: Drug Utilization and Quality of Life Study in Coronary Artery Disease Patients in a North Indian Tertiary Care Center
Brief Title: Drug Utilisation and Lifestyle Intervention Study in Patients Attending Cardiac Outpatient Clinic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KR Mangalam University (Other)
Responsible Party: Principal Investigator, Yojna Sah Jain, Research Scholar, KR Mangalam University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HappyHeartTrial
Record Dates: First submitted 2020-02-12; First posted 2020-02-17 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Early Intervention, Educational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Patients receiving an education program along with usual medical care
  Interventions: Behavioral: Education program
- Non Experimental (No Intervention): Patients receiving usual medical care

INTERVENTIONS:
Behavioral: Education program — A mobile application plus short message service (SMS) program to deliver disease-related health education and reinforcement to experimental group patients and see its impact on their health related quality of life, physical activity and Body mass index
  Arms: Experimental

SUMMARY:
This study has two parts: A drug utilization study and a Health-related quality of life study.

DETAILED DESCRIPTION:
This study has two parts: A drug utilization study and a Health-related quality of life study.

Drug utilisation study is an open label, cross sectional, descriptive drug utilization analysis of the primary cardiovascular drug classes prescribed to coronary artery disease patients attending cardiology OPD of a North India hospital.

Quality of life study intended to evaluate impact of a mobile based patient education program on the health related quality of life, physical activity and body mass index of coronary artery disease patients. It is a two arm study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults 18 - 75 years of age
* Diagnosed cased of coronary artery disease
* Agreeing after informed consent to participate

Exclusion Criteria:

* High risk cardiac patients
* Systemic, orthopedic and/or neurological problems restricting physical activity

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
HRQOL measured by RAND-Short form (SF)- 36 questionnaire | 9 months
  Health related quality of life to be measured using RAND-Short form (SF)- 36 questionnaire. This questionnaire comprises of 36 questions that measure HRQOL across 8 different domains that can be summarised into physical, mental and general health summary scores. Higher the SF 36 domain scores, better is the quality of life.

SECONDARY OUTCOMES:
Physical activity measured by International Physical Activity Questionnaire (IPAQ)- Short Form | 9 months
  Physical activity of the participants to be measured using International Physical Activity Questionnaire (IPAQ)- Short Form. It measures physical vigorous and moderate physical activity along with time spent in walking and sedentary activities. Higher the IPAQ score, higher is the physical activity.

OTHER OUTCOMES:
Body mass index | 9 months
  Body mass index for all patients

CONTACTS AND LOCATIONS:
Overall Officials: Yojna Jain, Masters, Principal Investigator — KR Mangalam University
Locations (1):
- Paras Hospital, Gurgaon, Haryana, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dibben G, Faulkner J, Oldridge N, Rees K, Thompson DR, Zwisler AD, Taylor RS. Exercise-based cardiac rehabilitation for coronary heart disease. Cochrane Database Syst Rev. 2021 Nov 6;11(11):CD001800. doi: 10.1002/14651858.CD001800.pub4. PMID 34741536